CLINICAL TRIAL: NCT02882854
Title: Guanfacine for PONV and Pain After Sinus Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Stephen Harvey, Assistant Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 160282
Record Dates: First submitted 2016-07-15; First posted 2016-08-30 (Estimated); Results first posted 2019-01-03 (Actual); Last update posted 2019-01-03 (Actual); Status verified 2018-12

CONDITIONS: Postoperative Nausea and Vomiting; Pain, Postoperative
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Pain, Postoperative | interventions — Guanfacine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Guanfacine (Experimental): Guanfacine 1 mg capsule by mouth, one time prior to surgery.
  Interventions: Drug: Guanfacine
- Placebo (Placebo Comparator): Placebo with a similar appearance to guanfacine by mouth one time prior to surgery
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Guanfacine — Patients will receive 1 mg of guanfacine to take orally.
  Arms: Guanfacine
Drug: Placebo — Patients will receive a placebo containing no drug that appears similarly to guanfacine to take orally.
  Arms: Placebo

SUMMARY:
Postoperative nausea and vomiting (PONV) and pain are the most common causes of Post Anesthesia Care Unit (PACU) discharge delay, with untreated PONV occurring in 20-30% of post-surgical patients. The effect of guanfacine (GF) administration on pain and nausea scores will be assessed with two groups. One group will receive 1 mg of GF to take orally and the other group will receive a similar appearing placebo (containing no drug) to take orally.

DETAILED DESCRIPTION:
Pain after surgery is commonly treated with narcotics which can potentiate PONV, further delaying PACU discharge. In multiple studies, alpha-2 agonists such as clonidine and dexmedetomidine reduce both the incidence of PONV and post-op pain, as well as requirements for postoperative analgesics. These actions are mediated via central alpha-2A receptors (A2AR). Of the A2AR agonists, guanfacine, though a weak antihypertensive agent, has the highest selectivity for the A2AR, but to date is untested for its potential to treat either PONV or post-operative pain.

ELIGIBILITY:
Inclusion Criteria:

* VUMC patients undergoing sinus surgery in MCE OR

Exclusion Criteria:

* Inability to read and freely consent
* Patients who take alpha-2 agonists routinely (guanfacine, clonidine, tizanidine)
* Patients undergoing sinus surgery planned for greater than 3 hours
* Patients with significant pre-existing pain, on chronic pain (opioid, methadone) therapy, severe fibromyalgia or other pre-existing pain condition in any body part
* Patients with preoperative nausea/vomiting at baseline.
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen T Harvey, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dolin SJ, Cashman JN, Bland JM. Effectiveness of acute postoperative pain management: I. Evidence from published data. Br J Anaesth. 2002 Sep;89(3):409-23. PMID 12402719
- [Background] Luttinger D, Ferrari R, Perrone MH, Haubrich DR. Pharmacological analysis of alpha-2 adrenergic mechanisms in nociception and ataxia. J Pharmacol Exp Ther. 1985 Mar;232(3):883-9. PMID 2857790
- [Background] Yamadera H, Ferber G, Matejcek M, Pokorny R. Electroencephalographic and psychometric assessment of the CNS effects of single doses of guanfacine hydrochloride (Estulic) and clonidine (Catapres). Neuropsychobiology. 1985;14(2):97-107. doi: 10.1159/000118212. PMID 3911096
- [Background] Connor DF, Arnsten AF, Pearson GS, Greco GF. Guanfacine extended release for the treatment of attention-deficit/hyperactivity disorder in children and adolescents. Expert Opin Pharmacother. 2014 Aug;15(11):1601-10. doi: 10.1517/14656566.2014.930437. Epub 2014 Jul 3. PMID 24992513
- [Background] Massad IM, Mohsen WA, Basha AS, Al-Zaben KR, Al-Mustafa MM, Alghanem SM. A balanced anesthesia with dexmedetomidine decreases postoperative nausea and vomiting after laparoscopic surgery. Saudi Med J. 2009 Dec;30(12):1537-41. PMID 19936416
- [Background] Kamibayashi T, Hayashi Y, Mammoto T, Yamatodani A, Sumikawa K, Yoshiya I. Role of the vagus nerve in the antidysrhythmic effect of dexmedetomidine on halothane/epinephrine dysrhythmias in dogs. Anesthesiology. 1995 Nov;83(5):992-9. doi: 10.1097/00000542-199511000-00013. PMID 7486186
- [Background] Unnerstall JR, Kopajtic TA, Kuhar MJ. Distribution of alpha 2 agonist binding sites in the rat and human central nervous system: analysis of some functional, anatomic correlates of the pharmacologic effects of clonidine and related adrenergic agents. Brain Res. 1984 Mar;319(1):69-101. doi: 10.1016/0165-0173(84)90030-4. PMID 6324960
- [Background] Giovannoni MP, Ghelardini C, Vergelli C, Dal Piaz V. Alpha2-agonists as analgesic agents. Med Res Rev. 2009 Mar;29(2):339-68. doi: 10.1002/med.20134. PMID 18680204
- [Background] Aghajanian GK, Wang YY. Common alpha 2- and opiate effector mechanisms in the locus coeruleus: intracellular studies in brain slices. Neuropharmacology. 1987 Jul;26(7B):793-9. doi: 10.1016/0028-3908(87)90054-2. PMID 2443865
- [Background] Ittermann T, Volzke H, Baumeister SE, Appel K, Grabe HJ. Diagnosed thyroid disorders are associated with depression and anxiety. Soc Psychiatry Psychiatr Epidemiol. 2015 Sep;50(9):1417-25. doi: 10.1007/s00127-015-1043-0. Epub 2015 Mar 17. PMID 25777685
- [Background] Baser E, Togrul C, Ozgu E, Esercan A, Caglar M, Gungor T. Effect of pre-procedural state-trait anxiety on pain perception and discomfort in women undergoing colposcopy for cervical cytological abnormalities. Asian Pac J Cancer Prev. 2013;14(7):4053-6. doi: 10.7314/apjcp.2013.14.7.4053. PMID 23991951
- [Background] Benarroch EE. The locus ceruleus norepinephrine system: functional organization and potential clinical significance. Neurology. 2009 Nov 17;73(20):1699-704. doi: 10.1212/WNL.0b013e3181c2937c. No abstract available. PMID 19917994
- [Background] Goldman-Rakic PS. Cellular basis of working memory. Neuron. 1995 Mar;14(3):477-85. doi: 10.1016/0896-6273(95)90304-6. No abstract available. PMID 7695894
- [Background] Wang M, Gamo NJ, Yang Y, Jin LE, Wang XJ, Laubach M, Mazer JA, Lee D, Arnsten AF. Neuronal basis of age-related working memory decline. Nature. 2011 Jul 27;476(7359):210-3. doi: 10.1038/nature10243. PMID 21796118
- [Background] Goldman-Rakic PS. Circuitry of the frontal association cortex and its relevance to dementia. Arch Gerontol Geriatr. 1987 Sep;6(3):299-309. doi: 10.1016/0167-4943(87)90029-x. PMID 3318747
- [Background] Hunt RD, Arnsten AF, Asbell MD. An open trial of guanfacine in the treatment of attention-deficit hyperactivity disorder. J Am Acad Child Adolesc Psychiatry. 1995 Jan;34(1):50-4. doi: 10.1097/00004583-199501000-00013. PMID 7860456
- [Background] Arnsten AF, Jin LE. Guanfacine for the treatment of cognitive disorders: a century of discoveries at Yale. Yale J Biol Med. 2012 Mar;85(1):45-58. Epub 2012 Mar 29. PMID 22461743
- [Background] Zhao X, Tong D, Long B, Wu X. [Effects of different doses of dexmedetomidine on the recovery quality from general anesthesia undergoing thyroidectomy]. Zhonghua Wei Zhong Bing Ji Jiu Yi Xue. 2014 Apr;26(4):239-43. doi: 10.3760/cma.j.issn.2095-4352.2014.04.008. Chinese. PMID 24709495
- [Background] Blaudszun G, Lysakowski C, Elia N, Tramer MR. Effect of perioperative systemic alpha2 agonists on postoperative morphine consumption and pain intensity: systematic review and meta-analysis of randomized controlled trials. Anesthesiology. 2012 Jun;116(6):1312-22. doi: 10.1097/ALN.0b013e31825681cb. PMID 22546966
- [Background] Lin TF, Yeh YC, Lin FS, Wang YP, Lin CJ, Sun WZ, Fan SZ. Effect of combining dexmedetomidine and morphine for intravenous patient-controlled analgesia. Br J Anaesth. 2009 Jan;102(1):117-22. doi: 10.1093/bja/aen320. Epub 2008 Nov 5. PMID 18987053
- [Background] Gurbet A, Basagan-Mogol E, Turker G, Ugun F, Kaya FN, Ozcan B. Intraoperative infusion of dexmedetomidine reduces perioperative analgesic requirements. Can J Anaesth. 2006 Jul;53(7):646-52. doi: 10.1007/BF03021622. PMID 16803911
- [Background] Ozkose Z, Demir FS, Pampal K, Yardim S. Hemodynamic and anesthetic advantages of dexmedetomidine, an alpha 2-agonist, for surgery in prone position. Tohoku J Exp Med. 2006 Oct;210(2):153-60. doi: 10.1620/tjem.210.153. PMID 17023769
- [Background] Tufanogullari B, White PF, Peixoto MP, Kianpour D, Lacour T, Griffin J, Skrivanek G, Macaluso A, Shah M, Provost DA. Dexmedetomidine infusion during laparoscopic bariatric surgery: the effect on recovery outcome variables. Anesth Analg. 2008 Jun;106(6):1741-8. doi: 10.1213/ane.0b013e318172c47c. PMID 18499604
- [Background] Rago R, Forfori F, Materazzi G, Abramo A, Collareta M, Miccoli P, Giunta F. Evaluation of a preoperative pain score in response to pressure as a marker of postoperative pain and drugs consumption in surgical thyroidectomy. Clin J Pain. 2012 Jun;28(5):382-6. doi: 10.1097/AJP.0b013e3182326495. PMID 22001665
- [Background] Hicks JA, Jenkins JG. The measurement of preoperative anxiety. J R Soc Med. 1988 Sep;81(9):517-9. doi: 10.1177/014107688808100907. PMID 3184108
- [Background] Charlson ME, Charlson RE, Peterson JC, Marinopoulos SS, Briggs WM, Hollenberg JP. The Charlson comorbidity index is adapted to predict costs of chronic disease in primary care patients. J Clin Epidemiol. 2008 Dec;61(12):1234-1240. doi: 10.1016/j.jclinepi.2008.01.006. Epub 2008 Jul 10. PMID 18619805
- [Background] Apfel CC, Laara E, Koivuranta M, Greim CA, Roewer N. A simplified risk score for predicting postoperative nausea and vomiting: conclusions from cross-validations between two centers. Anesthesiology. 1999 Sep;91(3):693-700. doi: 10.1097/00000542-199909000-00022. PMID 10485781
- [Background] Aubrun F, Langeron O, Quesnel C, Coriat P, Riou B. Relationships between measurement of pain using visual analog score and morphine requirements during postoperative intravenous morphine titration. Anesthesiology. 2003 Jun;98(6):1415-21. doi: 10.1097/00000542-200306000-00017. PMID 12766651

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Guanfacine | Placebo
Started | 40 | 44
Completed | 39 | 41
Not Completed | 1 | 3
Not completed — Lost to Follow-up | 1 | 2
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Guanfacine | Placebo | Total
Number analyzed (Participants) | 39 | 41 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 34 | 34 | 68
  >=65 years | 5 | 7 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (16.9) | 48.7 (15.4) | 45.3 (16.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 19 | 40
  Male | 18 | 22 | 40
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 39 | 41 | 80

OUTCOME MEASURES:

1. Primary Outcome: Comparison of PONV Score of Assessments Done at 15 Minutes After Arrival in PACU Using 11-point Nausea Scale (nVRS)
Description: Comparison of PONV Score of assessments done at 15 minutes after arrival in PACU using the nVRS when 0 is no nausea and 10 is worst nausea
Time Frame: 15 minutes after arriving in PACU
Population: 15 minute nVRS datapoint was not available for 2 participants in the Placebo group
Measure: Count of Participants; unit: Participants
Arm/Group | Guanfacine | Placebo
Number analyzed (Participants) | 39 | 39
Participants
  None (nVRS 0) | 35 | 33
  Mild (nVRS 1-5) | 1 | 2
  Moderate/Severe (nVRS 6-10) | 3 | 4

2. Primary Outcome: Comparison of PONV Score of Assessments Done at 30 Minutes After Arrival in PACU Using 11-point Nausea Scale (nVRS)
Description: Comparison of PONV Score of assessments done at 30 minutes after arrival in PACU using the nVRS when 0 is no nausea and 10 is worst nausea
Time Frame: 30 minutes after arriving in PACU
Measure: Count of Participants; unit: Participants
Arm/Group | Guanfacine | Placebo
Number analyzed (Participants) | 39 | 41
Participants
  None (nVRS 0) | 34 | 34
  Mild (nVRS 1-5) | 4 | 5
  Moderate/Severe (nVRS 6-10) | 1 | 2

3. Primary Outcome: Comparison of PONV Score of Assessments Done at 60 Minutes After Arrival in PACU Using 11-point Nausea Scale (nVRS)
Description: Comparison of PONV Score of assessments done at 60 minutes after arrival in PACU using the nVRS when 0 is no nausea and 10 is worst nausea
Time Frame: 60 minutes after arriving in PACU
Population: nVRS data was not available for 1 participant in the Guanfacine group
Measure: Count of Participants; unit: Participants
Arm/Group | Guanfacine | Placebo
Number analyzed (Participants) | 38 | 41
Participants
  None (nVRS 0) | 33 | 35
  Mild (nVRS 1-5) | 2 | 5
  Moderate/Severe (nVRS 6-10) | 3 | 1

4. Primary Outcome: Postoperative Nausea Assessment Using 11-point Nausea Scale (nVRS)
Description: PONV assessed using nVRS at 24 hours postop when 0 is no nausea and 10 is worst nausea.
Time Frame: 24 hours post op
Population: Only 70 patients (32 in guanfacine arm; 38 in placebo arm) responded to follow-up phone call and provided PONV data at the 24 hour timepoint.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Guanfacine | Placebo
Number analyzed (Participants) | 32 | 38
score on a scale | 0.00 [0.00 to 0.25] | 0.00 [0.00 to 0.00]

5. Secondary Outcome: Maximum Postoperative Pain Assessment Using 11-point Visual/Verbal Analog (VAS)
Description: Maximum postoperative pain assessment assessed in PACU at 15, 30 and 60 minutes after PACU arrival using VAS when 0 is no pain and 10 is worst pain
Time Frame: 15, 30, 60 minutes after arriving in PACU
Population: Data unavailable for 2 participants in the placebo group at 15 minute time point, 1 participant in the placebo group at the 30 minute time point,
Measure: Count of Participants; unit: Participants
Arm/Group | Guanfacine | Placebo
Number analyzed (Participants) | 39 | 41
Participants
  15 minutes after PACU admission: number analyzed (Participants) | 39 | 39
  15 minutes after PACU admission: None (Pain nVRS 0) | 31 | 24
  15 minutes after PACU admission: Mild (Pain nVRS 1-5) | 0 | 5
  15 minutes after PACU admission: Moderate/Severe (Pain nVRS 6-10) | 8 | 10
  30 minutes after PACU admission: number analyzed (Participants) | 39 | 40
  30 minutes after PACU admission: None (Pain nVRS 0) | 18 | 20
  30 minutes after PACU admission: Mild (Pain nVRS 1-5) | 7 | 6
  30 minutes after PACU admission: Moderate/Severe (Pain nVRS 6-10) | 14 | 14
  60 minutes after PACU admission: None (Pain nVRS 0) | 12 | 16
  60 minutes after PACU admission: Mild (Pain nVRS 1-5) | 6 | 13
  60 minutes after PACU admission: Moderate/Severe (Pain nVRS 6-10) | 21 | 12

6. Secondary Outcome: Postoperative Pain Assessment Using 11-point Visual/Verbal Analog (VAS)
Description: Postoperative pain assessment using VAS at 24 hours postop when 0 is no pain and 10 is worst pain
Time Frame: 24 hours postop
Population: Based on only 71 participants to post operative questionnaire.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Guanfacine | Placebo
Number analyzed (Participants) | 33 | 38
score on a scale | 3 [3 to 5] | 2 [1 to 4]

7. Secondary Outcome: Total Narcotic Requirement in PACU
Description: Total narcotic requirement in PACU tallied in morphine equivalents during PACU stay
Time Frame: Time frame between arrival and discharge in PACU, approximately 90 minutes
Population: Data was not available for 1 participant in the placebo group.
Measure: Median (Inter-Quartile Range); unit: morphine equivalents
Arm/Group | Guanfacine | Placebo
Number analyzed (Participants) | 39 | 40
morphine equivalents | 8.75 [4.38 to 18.88] | 7.50 [0.00 to 16.25]

8. Secondary Outcome: Number of Doses of PONV Treatment Administered in PACU
Time Frame: Time frame between arrival and discharge in PACU, approximately 90 minutes
Population: Data missing for1 participants in the placebo group and 1 participant in the Guanfacine group.
Measure: Count of Participants; unit: Participants
Arm/Group | Guanfacine | Placebo
Number analyzed (Participants) | 38 | 40
Participants
  Zero doses | 26 | 32
  One dose | 8 | 5
  Two doses | 4 | 3

9. Secondary Outcome: PACU Length of Stay in Minutes
Time Frame: Time frame between arrival and discharge in PACU, approximately 90 minutes
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Guanfacine | Placebo
Number analyzed (Participants) | 39 | 41
minutes | 128 [95 to 169.5] | 110 [87 to 155]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from consent to discharge from PACU (about 7 hours)
Arm/Group | Guanfacine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/44
Other Adverse Events (participants affected / at risk) | 0/40 | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-10): https://cdn.clinicaltrials.gov/large-docs/54/NCT02882854/Prot_SAP_000.pdf